CLINICAL TRIAL: NCT04028921
Title: Activity, Adiposity, and Appetite in Adolescents 2
Acronym: AAAA2
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Robin Shook, Associate Professor, Children's Mercy Hospital Kansas City
Other Study IDs: STUDY00001808; K01DK119545 (NIH)
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Metabolic Disease; Insulin Sensitivity
MeSH Terms: conditions — Obesity; Metabolic Diseases; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal weight, active: Male and female adolescents (age 14-17 years), BMI percentile >=5th to <75th for age/sex, >=60 min/day of moderate/vigorous physical activity.
  Interventions: Other: No intervention
- Normal weight, sedentary: Male and female adolescents (age 14-17 years), BMI percentile >=5th to <75th for age/sex, <60 min/day of moderate/vigorous physical activity.
  Interventions: Other: No intervention
- Overweight/obese, active: Male and female adolescents (age 14-17 years), BMI percentile >=85th to <99th for age/sex, >=60 min/day of moderate/vigorous physical activity.
  Interventions: Other: No intervention
- Overweight/obese, sedentary: Male and female adolescents (age 14-17 years), BMI percentile >=85th to <99th for age/sex, <60 min/day of moderate/vigorous physical activity.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a cross-sectional study; no intervention

SUMMARY:
Our goal is to examine linkages between physical activity, appetite control, and energy metabolism in adolescents. The investigators will assess metabolic function and appetite control in male and female adolescents stratified by bodyweight and physical activity using across-sectional study design.

DETAILED DESCRIPTION:
Childhood obesity is the most serious public health problem of the 21st century, given the prevalence, global reach, and widespread health, economic, and social consequences. While weight gain at the most basic level is due to a chronic energy surplus, there are a host of influences that act on the energy balance system that remain largely unknown. Thus, there is a critical need to identify previously unexamined factors that may influence the energy balance system in order to develop effective interventions for prevention and treatment. Our long-term goal is to quantify the dynamic relationships between various physiological and psychological components of the energy balance system. Our short-term goal is to examine linkages between physical activity, appetite control, and energy metabolism in adolescents. The status quo as it relates to appetite control is that body weight status and related peripheral signals are a key regulator of energy intake. In contrast to body weight playing a primary role in energy regulation, our working hypothesis is that high levels of regular moderate-to-vigorous physical activity (MVPA) result in a metabolic phenotype consisting of enhanced metabolic function and proper regulation of appetite, which prevents the development of obesity. The investigators have reported that adults with low levels of MVPA have dysregulated appetite control, evidenced by higher levels of energy intake and elevated levels of dietary disinhibition. Additionally, the investigators have observed that rats with low fitness possess dysregulated control of appetite and reduced hepatic fat oxidation compared to rats with high fitness. Based on these findings in adults and rodents, in addition to supportive work by others, the investigators hypothesize that low levels of MVPA create a metabolic phenotype, leading to dysregulated appetite control which predisposes individuals to weight gain. To test this hypothesis the investigators will perform a study focused on the links between physical activity and appetite. The investigators will assess metabolic function and appetite control in male and female adolescents stratified by bodyweight (normal vs overweight/obese) and physical activity (sedentary vs. active) using a 2 x 2 cross-sectional study design (N=44). The specific aim of the proposed study is: 1) To examine the association between physical activity and appetite control in adolescents, with metabolic function serving as a mediator. At the completion of the study, it is our expectation that the investigators will have described the independent effects of physical activity and body weight on energy metabolism and appetite in adolescents. This study will have a significant positive impact on the understanding of energy balance in adolescents, and will inform public health interventions that specifically target mechanisms associated with weight gain in youth.

ELIGIBILITY:
Inclusion Criteria:

* Tanner Stage III-V
* Non-smoking
* Not currently involved in any other research study

Exclusion Criteria:

* Restrained eater (>13) on the restraint section of the three-factor eating questionnaire; Current/past diagnosis of an eating disorder
* Gave birth in the past 12 months or <6 months post-lactation.
* Self-reported medical conditions (diabetes, Crohn's disease, etc.) that may affect adherence to the protocol or exercising safely or alter metabolism
* Medications known to affect exercise performance or metabolism (e.g. thyroid medication, beta-blockers, or stimulants)

Ages: 14 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Healthy males and females.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin P Shook, PhD, Principal Investigator — Children's Mercy
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Aggregated results will be shared

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Weight, Active | Normal Weight, Sedentary | Overweight/Obese, Active | Overweight/Obese, Sedentary
Started | 13 | 11 | 12 | 10
Completed | 13 | 11 | 12 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Weight, Active | Normal Weight, Sedentary | Overweight/Obese, Active | Overweight/Obese, Sedentary | Total
Number analyzed (Participants) | 13 | 11 | 12 | 10 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 11 | 12 | 10 | 46
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.9 (0.3) | 16.0 (0.4) | 16.4 (0.4) | 16.4 (0.4) | 16.0 (0.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 8 | 6 | 31
  Male | 6 | 1 | 4 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 4 | 0 | 9
  Not Hispanic or Latino | 11 | 8 | 8 | 10 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 1 | 5 | 11
  White | 10 | 8 | 11 | 5 | 34
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 11 | 12 | 10 | 46

OUTCOME MEASURES:

1. Primary Outcome: Appetite- Subjective
Description: The investigators will measure subjective appetite ratings using visual analog scales related to hunger following a fixed-calorie meal: Hunger, Area Under the Curve (AUC)
  Hunger and palatability were assessed using self-rated visual analogue scales (Rogers, P. J., & Blundell, J. E. (1993). Intense sweeteners and appetite. The American Journal of Clinical Nutrition, 58(1), 120-122.) Scale is 0-100, with 0 equaling 'I am not hungry at all' and 100 equaling 'I have never been more hungry'.
  Area under the curve (AUC) was calculated for appetite variables by calculating the area of the response as you would a trapezoid.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale*min
Arm/Group | Normal Weight, Active | Normal Weight, Sedentary | Overweight/Obese, Active | Overweight/Obese, Sedentary
Number analyzed (Participants) | 13 | 11 | 12 | 10
score on a scale*min | 9239.4 (3635.1) | 7879.6 (5343.5) | 6130.5 (4279.7) | 8970.0 (3664.9)

2. Primary Outcome: Appetite- Objective
Description: The investigators will measure objective appetite responses using plasma ghrelin following a fixed-calorie meal.
Time Frame: Baseline
Population: Plasma ghrelin values were not assessed. Blood samples needed for assessment were not obtained due to lack of staff. Samples will not be collected in the future.
Arm/Group | Normal Weight, Active | Normal Weight, Sedentary | Overweight/Obese, Active | Overweight/Obese, Sedentary
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Primary Outcome: Appetite- Adjusted
Description: The investigators will measure objective and subjective appetite responses as described above adjusted by insulin sensitivity (glucose infusion rate, mg/kg/min) as assessed in the euglycemic hyperinsulinemic clamp technique.
  Hunger score on a scale*min adjusted for glucose infusion rate (mL/kgFFM/min) and sex
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale*min
Arm/Group | Normal Weight, Active | Normal Weight, Sedentary | Overweight/Obese, Active | Overweight/Obese, Sedentary
Number analyzed (Participants) | 13 | 11 | 12 | 10
score on a scale*min | 8686 (1414) | 7885 (1442) | 6534 (1528) | 8703 (1537)

ADVERSE EVENTS:
Time Frame: Baseline
Arm/Group | Normal Weight, Active | Normal Weight, Sedentary | Overweight/Obese, Active | Overweight/Obese, Sedentary
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 2/13 | 2/11 | 2/12 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Weight, Active (N=13) | Normal Weight, Sedentary (N=11) | Overweight/Obese, Active (N=12) | Overweight/Obese, Sedentary (N=10)
Extravasation of IV (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lightheadedness during IV placement (Vascular disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT04028921/Prot_SAP_000.pdf